CLINICAL TRIAL: NCT00915772
Title: Extension Study Linagliptin 2.5 mg Bid + Metformin 500 or 1000 mg Bid Versus Metformin 1000 mg Bid
Brief Title: Treatment of Type 2 Diabetes With Linagliptin 2.5 mg Bid + Metformin 500 or 1000 mg Bid and Metformin 1000 mg Bid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.52; 2008-008494-59 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-06-02; First posted 2009-06-08 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Metformin

ARMS (3):
- Linagliptin + metformin bid (Experimental): Linagliptin low dose + metformin 500 mg, bid
  Interventions: Drug: Linagliptin + metformin
- Linagliptin+ metformin bid (Experimental): Linagliptin low dose + metformin 1000 mg bid
  Interventions: Drug: Linagliptin+metformin
- Metformin bid (Active Comparator): Metformin 1000 mg bid
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Linagliptin + metformin — Linagliptin tablet low dose + metformin tablet 500 mg bid
  Arms: Linagliptin + metformin bid
Drug: Linagliptin+metformin — Linagliptin low dose tablet + metformin 1000 mg tablet bid
  Arms: Linagliptin+ metformin bid
Drug: Metformin — Metformin 1000 mg tablet bid
  Arms: Metformin bid

SUMMARY:
A phase III randomised, double-blind parallel group extension study to investigate the efficacy and safety of twice daily administration of the free combination of linagliptin 2.5 mg + metformin 500 mg or of linagliptin 2.5 mg + metformin 1000 mg versus monotherapy with metformin 1000 mg twice daily over 54 weeks in type 2 diabetic patients previously completing the double-blind part of study 1218.46

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent, at the latest by the date of Visit 1
* Patients completing the entire treatment period of the double-blind study 1218.46, who are not treated with rescue medication (Visit 7)

Exclusion criteria:

* Patients who meet one or more of the withdrawal criteria of the treatment period of the previous study 1218.46
* Pre-menopausal women (last menstruation equal or less than 1 year prior to signing informed consent) who:
* are nursing or pregnant,
* or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner and in addition for male partners a barrier method, such as the use of condom with spermicide. No exception will be made.
* Alcohol abuse within the 3 months prior to informed consent that would interfere with study participation
* Drug abuse that in the opinion of the investigator would interfere with trial participation
* Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (112):
- Canada (8):
  - 1218.52.11005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.52.11003 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1218.52.11002 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1218.52.11006 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.52.11008 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1218.52.11004 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.52.11007 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1218.52.11010 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Croatia (5):
  - 1218.52.38502 Boehringer Ingelheim Investigational Site, Karlovac
  - 1218.52.38503 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1218.52.38504 Boehringer Ingelheim Investigational Site, Osijek
  - 1218.52.38505 Boehringer Ingelheim Investigational Site, Rijeka
  - 1218.52.38501 Boehringer Ingelheim Investigational Site, Sisak
- Estonia (3):
  - 1218.52.37202 Boehringer Ingelheim Investigational Site, Pärnu
  - 1218.52.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1218.52.37203 Boehringer Ingelheim Investigational Site, Tallinn
- France (25):
  - 1218.52.3303D Boehringer Ingelheim Investigational Site, Aire Sur l'Aadour
  - 1218.52.3308B Boehringer Ingelheim Investigational Site, Bischheim
  - 1218.52.3305A Boehringer Ingelheim Investigational Site, Bourges
  - 1218.52.3304F Boehringer Ingelheim Investigational Site, Bousse
  - 1218.52.3308C Boehringer Ingelheim Investigational Site, Gambsheim
  - 1218.52.3301A Boehringer Ingelheim Investigational Site, Grenoble Cédex
  - 1218.52.3305B Boehringer Ingelheim Investigational Site, Guérigny
  - 1218.52.3304A Boehringer Ingelheim Investigational Site, Jarny
  - 1218.52.3302D Boehringer Ingelheim Investigational Site, La Riche
  - 1218.52.9999 Boehringer Ingelheim Investigational Site, La Riche
  - 1218.52.3307A Boehringer Ingelheim Investigational Site, La Seyne-sur-Mer
  - 1218.52.3307E Boehringer Ingelheim Investigational Site, La Seyne-sur-Mer
  - 1218.52.3305G Boehringer Ingelheim Investigational Site, Lury-sur-Arnon
  - 1218.52.3303A Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1218.52.3308F Boehringer Ingelheim Investigational Site, Mundolsheim
  - 1218.52.3305E Boehringer Ingelheim Investigational Site, Nevers
  - 1218.52.3306A Boehringer Ingelheim Investigational Site, Orthez
  - 1218.52.3306C Boehringer Ingelheim Investigational Site, Orthez
  - 1218.52.3303B Boehringer Ingelheim Investigational Site, Saint-Martin-d'Oney
  - 1218.52.3302E Boehringer Ingelheim Investigational Site, Savonnières
  - 1218.52.3308A Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.52.3308D Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.52.3308E Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.52.3307D Boehringer Ingelheim Investigational Site, Toulon
  - 1218.52.3302A Boehringer Ingelheim Investigational Site, Tours
- Germany (4):
  - 1218.52.49002 Boehringer Ingelheim Investigational Site, Bad Dürrheim-Sunthausen
  - 1218.52.49006 Boehringer Ingelheim Investigational Site, Cologne
  - 1218.52.49003 Boehringer Ingelheim Investigational Site, München
  - 1218.52.49007 Boehringer Ingelheim Investigational Site, Schauenburg
- India (18):
  - 1218.52.91009 Boehringer Ingelheim Investigational Site, Aurangabad
  - 1218.52.91001 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.52.91004 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.52.91012 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.52.91011 Boehringer Ingelheim Investigational Site, Bhopal
  - 1218.52.91003 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.52.91020 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.52.91018 Boehringer Ingelheim Investigational Site, Hyderadad
  - 1218.52.91008 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.52.91002 Boehringer Ingelheim Investigational Site, Karnataka
  - 1218.52.91007 Boehringer Ingelheim Investigational Site, Karnataka
  - 1218.52.91019 Boehringer Ingelheim Investigational Site, Madurai
  - 1218.52.91013 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.52.91015 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.52.91014 Boehringer Ingelheim Investigational Site, Nagpru
  - 1218.52.91016 Boehringer Ingelheim Investigational Site, P.O.Trivandrum
  - 1218.52.91010 Boehringer Ingelheim Investigational Site, Pune
  - 1218.52.91006 Boehringer Ingelheim Investigational Site, West Bengal
- Lithuania (3):
  - 1218.52.37001 Boehringer Ingelheim Investigational Site, Kaunas
  - 1218.52.37004 Boehringer Ingelheim Investigational Site, Kaunas
  - 1218.52.37003 Boehringer Ingelheim Investigational Site, Vilnius
- Mexico (7):
  - 1218.52.52006 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1218.52.52002 Boehringer Ingelheim Investigational Site, Cuernavaca
  - 1218.52.52004 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.52.52007 Boehringer Ingelheim Investigational Site, México
  - 1218.52.52008 Boehringer Ingelheim Investigational Site, México
  - 1218.52.52010 Boehringer Ingelheim Investigational Site, Tijuana
  - 1218.52.52009 Boehringer Ingelheim Investigational Site, Veracruz
- Netherlands (8):
  - 1218.52.31004 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.52.31005 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.52.31001 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1218.52.31002 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1218.52.31010 Boehringer Ingelheim Investigational Site, Breda
  - 1218.52.31013 Boehringer Ingelheim Investigational Site, Groningen
  - 1218.52.31014 Boehringer Ingelheim Investigational Site, Velp
  - 1218.52.31015 Boehringer Ingelheim Investigational Site, Zoetermeer
- Romania (5):
  - 1218.52.40001 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1218.52.40005 Boehringer Ingelheim Investigational Site, Galati
  - 1218.52.40003 Boehringer Ingelheim Investigational Site, Oradea
  - 1218.52.40002 Boehringer Ingelheim Investigational Site, Ploieşti
  - 1218.52.40004 Boehringer Ingelheim Investigational Site, Satu Mare
- Russia (7):
  - 1218.52.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.52.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.52.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.52.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.52.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.52.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.52.70007 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Sweden (4):
  - 1218.52.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.52.46003 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.52.46005 Boehringer Ingelheim Investigational Site, Stockholm
  - 1218.52.46001 Boehringer Ingelheim Investigational Site, Uppsala
- Tunisia (9):
  - 1218.52.2162A Boehringer Ingelheim Investigational Site, Bab Saâdoun Tunis
  - 1218.52.2162B Boehringer Ingelheim Investigational Site, Bab Sâadoun Tunis
  - 1218.52.9992 Boehringer Ingelheim Investigational Site, Bab Sâadoun Tunis
  - 1218.52.2161A Boehringer Ingelheim Investigational Site, Tunis
  - 1218.52.2161B Boehringer Ingelheim Investigational Site, Tunis
  - 1218.52.2163A Boehringer Ingelheim Investigational Site, Tunis
  - 1218.52.2163B Boehringer Ingelheim Investigational Site, Tunis
  - 1218.52.9991 Boehringer Ingelheim Investigational Site, Tunis
  - 1218.52.9993 Boehringer Ingelheim Investigational Site, Tunis
- Ukraine (6):
  - 1218.52.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.52.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.52.38005 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.52.38002 Boehringer Ingelheim Investigational Site, Odesa
  - 1218.52.38004 Boehringer Ingelheim Investigational Site, Odesa
  - 1218.52.38006 Boehringer Ingelheim Investigational Site, Vinnitsa

REFERENCES:
- See also: List of publications — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1218/1218.52_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 567 patients were entered and randomised, but only 566 were treated. Therefore the treated set (TS) comprises 566 patients.
Groups:
- M1000: Metformin 1000mg monotherapy twice daily
- L2.5+M500: Linagliptin 2.5mg and metformin 500mg twice daily
- L2.5+M1000: Linagliptin 2.5mg and metformin 1000mg twice daily
Period: Overall Study
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Started | 170 | 225 | 171
Completed | 134 | 179 | 142
Not Completed | 36 | 46 | 29
Not completed — Adverse Event | 12 | 13 | 11
Not completed — Protocol Violation | 4 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Lack of Efficacy | 9 | 15 | 3
Not completed — Refused to continue trial medication | 6 | 8 | 4
Not completed — Any other reason | 4 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000 | Total
Number analyzed (Participants) | 170 | 225 | 171 | 566
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (10.7) | 56.0 (10.7) | 55.7 (10.8) | 55.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 105 | 74 | 256
  Male | 93 | 120 | 97 | 310
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m2] | 29.33 (5.22) | 29.06 (4.95) | 28.64 (4.79) | 29.01 (4.98)
Baseline weight [Mean (Standard Deviation); unit: kg] | 81.09 (18.92) | 79.17 (18.75) | 78.62 (16.86) | 79.58 (18.25)
Baseline Glycosylated haemoglobin (HbA1c) at baseline [Mean (Standard Deviation); unit: percent] — Based upon non-missing data, n=559 (5:1:1 missing in each of the groups respectively)
  percent | 7.48 (0.99) | 7.64 (1.04) | 7.35 (1.12) | 7.50 (1.06)
Fasting plasma glucose (FPG) at baseline [Mean (Standard Deviation); unit: mg/dL] — Based upon non-missing data, n=544 (6:10:6 missing in each of the groups respectively)
  mg/dL | 156.585 (39.194) | 167.088 (44.633) | 153.721 (37.128) | 159.868 (41.206)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Patients With Adverse Events (AEs)
Description: This includes any AEs detected during routine physical examination and electrocardiogram (ECG) procedures.
Time Frame: 54 weeks
Population: Treated Set (TS): all screened patients who were documented to have taken at lease 1 dose of study drug.
Measure: Number; unit: participant
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 170 | 225 | 171
participant
  Patients with any AEs | 124 | 149 | 132
  Patients with severe AEs | 4 | 7 | 5
  Patients with withdrawal due to AEs (from AE page) | 10 | 11 | 9

2. Primary Outcome: Change From Baseline at Week 54 in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Baseline is defined as Visit 1 of 1218.52.
Time Frame: 54 weeks
Population: TS and observed cases (OC)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 164 | 214 | 165
mmHg
  DBP change from baseline | -0.3 (8.5) | -0.1 (7.4) | 0.3 (8.8)
  SBP change from baseline | 0.6 (12.2) | -0.2 (13.2) | 2.2 (13.6)

3. Primary Outcome: Change From Baseline at Week 54 in Pulse Rate
Description: Baseline is defined as Visit 1 of 1218.52.
Time Frame: 54 weeks
Population: TS and observed cases (OC)
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 164 | 214 | 164
beats per minute (bpm) | 0.0 (7.7) | 0.6 (8.3) | 0.1 (8.3)

4. Primary Outcome: Frequency of Patients With Possibly Clinically Significant Abnormal Laboratory Parameters: Haematology
Time Frame: 54 weeks
Population: TS and observed cases (OC)
Measure: Number; unit: participants
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 168 | 225 | 170
participants
  Haematocrit abnormality: <=32% | 2 | 2 | 0
  Haemoglobin abnormality:Female ≤9.5;Male ≤11.5g/dL | 7 | 4 | 2
  Red Blood Cells abnormality: < 3* 10^12/L | 0 | 0 | 0
  White Blood Cells abnormal decrease: < 3 * 10^9/L | 0 | 3 | 1
  White Blood Cells abnormal increase: <20.1*10^9/L | 0 | 1 | 0
  Platelets abnormal decrease: <= 75* 10^9/L | 0 | 0 | 1
  Platelets abnormal increase: >= 700* 10^9/L | 0 | 0 | 0

5. Primary Outcome: Possibly Clinically Significant Abnormal Laboratory Parameters: Clinical Chemistry
Description: ULN means upper limit of normal
Time Frame: 54 weeks
Population: TS and observed cases (OC). In treatment group L2.5+M500, the number of patients analysed was 224 for lactate dehydrogenase abnormality and total bilirubin abnormality due to anailable data.
Measure: Number; unit: participants
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 168 | 225 | 171
participants
  Eosinophils abnormality : ≥ 10% | 2 | 4 | 6
  Sodium abnormal decrease: < 130 mmol/L | 0 | 1 | 2
  Sodium abnormal increase: > 160 mmol/L | 1 | 0 | 0
  Potassium abnormal decrease: < 3 mmol/L | 0 | 0 | 0
  Potassium abnormal increase: > 5.8 mmol/L | 2 | 2 | 4
  Calcium abnormal decrease: < 1.8 mmol/L | 2 | 1 | 0
  Calcium abnormal increase: > 3 mmol/L | 0 | 1 | 0
  Phosphate abnormal decrease: < 0.7 mmol/L | 1 | 0 | 0
  Phosphate abnormal increase: > 1.7 mmol/L | 0 | 2 | 1
  Aspartate Transaminase abnormality: ≥3xULN | 3 | 2 | 2
  Alanine Transaminase (ALT) abnormality: >= 3 x ULN | 4 | 3 | 2
  Alkaline phosphatase abnormality: >= 2 x ULN | 1 | 0 | 0
  γ-glutamyl transpeptidase (GGT) increase:≥3ULN | 8 | 5 | 7
  Lactate dehydrogenase abnormality: >= 3 x ULN | 0 | 0 | 0
  Creatine kinase abnormality: >= 3 x ULN | 3 | 1 | 2
  Amylase: > 1.5 x ULN | 2 | 5 | 4
  Total cholesterol abnormality: > 300 mg/dL | 0 | 0 | 1
  Creatinine abnormality: >= 1.5 mg/dL | 0 | 1 | 0
  Total bilirubin abnormality: >= 2 mg/dL | 0 | 1 | 0
  Triglyceride abnormality: >300 mg/dL | 14 | 14 | 10
  Uric acid abnormality:Female: >10;Male: >11 mg/dL | 4 | 3 | 6
  Albumin abnormality: <2.5 g/dL | 0 | 1 | 0
  Bicarbonate abnormal decrease: <21 mmol/L | 0 | 0 | 2

6. Secondary Outcome: Change in HbA1c From Baseline Over Time
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the visit HbA1c percent minus the baseline HbA1c percent. Baseline is defined as visit 1 of 1218.52.
Time Frame: 54 weeks
Population: TS (OC) with non-missing data at visit
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 168 | 225 | 171
Percentage
  Change in HbA1c to week 6 (n=157, 207 and 166) | -0.06 (0.41) | -0.24 (0.51) | -0.26 (0.59)
  Change in HbA1c to week 18 (n=136, 184 and 147) | -0.08 (0.56) | -0.29 (0.79) | -0.34 (0.93)
  Change in HbA1c to week 30 (n=121, 165 and 134) | -0.10 (0.82) | -0.41 (0.80) | -0.36 (0.87)
  Change in HbA1c to week 42 (n=110, 152 and 127) | -0.14 (0.78) | -0.35 (0.80) | -0.28 (1.00)
  Change in HbA1c to week 54 (n=98, 132 and 117) | -0.06 (0.77) | -0.28 (0.86) | -0.24 (0.91)

7. Secondary Outcome: Number of Patients With HbA1c <7.0% After 54 Weeks
Time Frame: 54 weeks
Population: Treated Set with non completers considered as failures (NCF)
Measure: Number; unit: participant
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 170 | 225 | 171
participant
  No | 119 | 168 | 104
  Yes | 51 | 57 | 67

8. Secondary Outcome: Number of Patients With HbA1c <6.5% Over Time
Time Frame: 54 weeks
Population: Treated Set with non completers considered as failures (NCF)
Measure: Number; unit: participant
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 170 | 225 | 171
participant
  No | 148 | 196 | 130
  Yes | 22 | 29 | 41

9. Secondary Outcome: Number of Patients With HbA1c of at Least <0.5% Over Time
Time Frame: 54 weeks
Population: Treated Set with non completers considered as failures (NCF)
Measure: Number; unit: participant
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 170 | 225 | 171
participant
  No | 143 | 176 | 135
  Yes | 27 | 49 | 36

10. Secondary Outcome: Change in FPG From Baseline Over Time
Description: Baseline is defined as visit 1 of 1218.52.
Time Frame: 54 weeks
Population: TS (OC) with non-missing data at visit
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 168 | 225 | 171
mg/dL
  Change in FPG to week 2 (n=158, 200 and 158) | -4.36 (27.86) | -12.22 (28.70) | -10.57 (28.15)
  Change in FPG to week 6 (n=152, 189 and 157) | -4.18 (32.68) | -13.28 (27.36) | -13.46 (32.97)
  Change in FPG to week 18 (n=133, 174 and 142) | -1.14 (43.18) | -11.76 (33.10) | -12.88 (33.74)
  Change in FPG to week 30 (n=116, 156 and 130) | -7.22 (41.67) | -13.49 (33.68) | -13.90 (32.07)
  Change in FPG to week 42 (n=103, 149 and 124) | -7.43 (30.48) | -9.46 (33.61) | -13.10 (34.96)
  Change in FPG to week 54 (n=93, 132 and 115) | -6.02 (29.25) | -7.24 (36.27) | -9.82 (31.83)

11. Secondary Outcome: Number of Patients With Rescue Therapy
Time Frame: 54 weeks
Population: TS
Measure: Number; unit: Number of patients
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 170 | 225 | 171
Number of patients
  No | 128 | 163 | 147
  Yes | 42 | 62 | 24

12. Secondary Outcome: Change in HbA1c From Baseline Over Time
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the visit HbA1c percent minus the baseline HbA1c percent. Baseline is defined as visit 3 from study 1218.46 (NCT00915772).
Time Frame: 78 weeks
Population: Non-switcher set (OC) with non-missing data at visit. Only patients who continued on the same treatment in both studies are included
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Number analyzed (Participants) | 109 | 113 | 111
Percentage
  Change in HbA1c to week 30 (n=102, 103 and 108) | -1.19 (0.98) | -1.34 (0.91) | -1.74 (0.98)
  Change in HbA1c to week 42 (n=90, 92 and 95) | -1.16 (0.98) | -1.31 (0.99) | -1.62 (1.05)
  Change in HbA1c to week 54 (n=81, 81 and 87) | -1.20 (1.14) | -1.41 (1.03) | -1.73 (0.99)
  Change in HbA1c to week 66 (n=74, 73 and 84) | -1.26 (1.02) | -1.42 (0.93) | -1.65 (1.09)
  Change in HbA1c to week 78 (n=66, 66 and 78) | -1.25 (0.91) | -1.32 (1.06) | -1.63 (1.05)

13. Primary Outcome: Clinical Relevant Drug-related Abnormal Findings in Physical Examination and ECG as Reported as AE
Description: Frequency of patients with adverse events by treatment, primary system organ class and preferred term
Time Frame: Baseline and drug stop (up to 54 weeks) + 7 days
Population: Treated Set (TS)
Measure: Number; unit: participants
Groups:
- Post-treat: 7 days follow-up period
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000 | Post-treat
Number analyzed (Participants) | 170 | 225 | 171 | 566
participants
  Cardiogenic shock | 0 | 0 | 1 | 0
  Supraventricular tachycardia | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 54 weeks
Groups:
- M1000: Metformin 1000 mg twice daily
- L2.5+M500: Linagliptin 2.5 mg + Metformin 500 mg twice daily
- L2.5+M1000: Linagliptin 2.5 mg + Metformin 1000 mg twice daily
Arm/Group | M1000 | L2.5+M500 | L2.5+M1000
Serious Adverse Events (participants affected / at risk) | 7/170 | 12/225 | 14/171
Other Adverse Events (participants affected / at risk) | 63/170 | 87/225 | 77/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M1000 (N=170) | L2.5+M500 (N=225) | L2.5+M1000 (N=171)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Holoprosencephaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M1000 (N=170) | L2.5+M500 (N=225) | L2.5+M1000 (N=171)
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 12
Nasopharyngitis (Infections and infestations) | 9 | 9 | 12
Urinary tract infection (Infections and infestations) | 4 | 9 | 9
Glomerular filtration rate decreased (Investigations) | 6 | 14 | 11
Glycosylated haemoglobin increased (Investigations) | 9 | 12 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 14 | 18 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 29 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 11 | 11
Hypertension (Vascular disorders) | 9 | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.